CLINICAL TRIAL: NCT03881397
Title: Youth Health and Social Media: Objective 2 Pilot Intervention
Brief Title: Youth Health and Social Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Facebook, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-0787; A536760 (Other: UW, Madison); SMPH/PEDIATRICS/GPAM (Other: UW, Madison)
Record Dates: First submitted 2018-06-21; First posted 2019-03-19 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Sleep; Physical Activity; Family and Household; Computer, Attitude to; Adolescent Behavior
Keywords: internet; social media; family rules
MeSH Terms: conditions — Motor Activity; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Track A will be our intervention group receiving the Family Media Use intervention Track B will serve as control group at Time 2, and then receive an awareness intervention at that time to compare that intervention at Time 3 to Track A at Time 2
Masking Description: This will be an online intervention with interventions pre-determined by tracks, so no masking is needed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Track B assessed at Time 2) (No Intervention): A survey regarding tech use, health behaviors and well-being including physical activity, anxiety, and sleep
- Online Family Media Use Plan (Track A) (Experimental): The Online Family Media Use Plan group will receive a link to American Academy of Pediatrics Family Media Use plan at the end of the survey, which describes internet safety ideas for teens and parents to review and create together.
  Interventions: Behavioral: Family Media Use Plan
- Media Use Resources Awareness (Track B assessed at Time 3) (Experimental): Resources offered to parents and teens that include tools and data for safe technology use among teens
  Interventions: Behavioral: Media Use Resources Awareness

INTERVENTIONS:
Behavioral: Family Media Use Plan — A tool developed by the American Academy of Pediatrics that engages teens and parent to discuss internet safety ideas and develop rules around technology use together.
  Arms: Online Family Media Use Plan (Track A)
Behavioral: Media Use Resources Awareness — Resources offered to parents and teens that include tools and publicly available resources for safe technology use among teens
  Arms: Media Use Resources Awareness (Track B assessed at Time 3)

SUMMARY:
The purpose of this study is test the American Academy of Pediatrics (AAP) Family Media Use plan among teens and their parents through a randomized intervention and assess impact on outcomes including family media rules and health behavior outcomes.

DETAILED DESCRIPTION:
For this study there will be three time points of data collection and participant contact by Qualtrics:

Time 1: Baseline

Participants (teen and parent dyads) will be randomized into one of two tracks:

Track A: Family Media Use Plan intervention Track B: Awareness intervention (delayed start intervention)

The track A group will complete a survey regarding technology rules, tech use, and health behaviors, as well as the Family Media Use Plan embedded into the survey. Track B group will only complete the baseline survey.

Time 2: Follow Up Survey: 4-6 weeks after baseline

Track A group will complete a follow-up survey similar to the baseline with additional follow-up questions around their use of the family media use plan.

The track B group will complete a similar survey and receive the Awareness Intervention, providing resources available regarding youth and media use .

Time 3: Follow Up Survey: 3-4 months after baseline

All participants will be asked to complete their corresponding tracks (track A or track B) survey again to understand use media use and health behaviors change over time.

Track A or B designated questions are labeled within each uploaded survey.

ELIGIBILITY:
Inclusion Criteria:

* English speaking and between the ages of 12 and 17
* Parents must be English speaking and have a child between the ages of 12 and 17

Exclusion Criteria:

* n/a

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1520 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Technology and Media Use Rules | 4 months after initial baseline
  Increases in the number of positive responses to technology and media rules followed or maintained

SECONDARY OUTCOMES:
Changes in sleep behavior | 2 and 4 months after initial baseline (Time 2 and 3)
  Changes in sleep as measured by the 8 item Pediatric Daytime Sleepiness Scale (PDSS). Participants will assess their sleep behaviors by answering each item with "never", "seldom", "sometimes", "frequently", or "always". Items are scored from 0-4 (never= 0; seldom=1; sometimes=2; frequently=3; always=4) with a score above 16 indicating poor sleep behavior.
Changes in risk for Problematic Internet Use | 2 and 4 months after initial baseline (Time 2 and 3)
  Changes in problematic internet use symptoms as measured by the 18-item Problematic and Risky Internet Use Screening Scale (PRIUSS). For each item participants will select from "never", "rarely", "sometimes", "often", or "very often" in relation to their internet use over the last 6 months. Each option is coded with "never" equal to 1 and "very often" equal to 5. An overall composite score is calculated at the end, with an overall score of 25 indicating a risk for problematic internet use.

OTHER OUTCOMES:
Changes in physical activity | 2 and 4 months after initial baseline (Time 2 and 3)
  Reported physical activity as measured by the 3 item Physical Activity Scale. Response options range from never (1) to 4 times or more a week (5) for each item. Higher scores indicating greater physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Moreno, MD, MPH, MSeD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moreno MA, Binger KS, Zhao Q, Eickhoff JC. Effect of a Family Media Use Plan on Media Rule Engagement Among Adolescents: A Randomized Clinical Trial. JAMA Pediatr. 2021 Apr 1;175(4):351-358. doi: 10.1001/jamapediatrics.2020.5629. PMID 33492346